CLINICAL TRIAL: NCT02457039
Title: An Assessor-Blinded, Randomised Controlled Trial of Acupuncture to Prevent Chemobrain in Breast Cancer Patients
Brief Title: Acupuncture Prevents Chemobrain in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Zhang Zhang-Jin, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UW 14-206
Record Dates: First submitted 2015-05-15; First posted 2015-05-29 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Chemo-brain; Drug-Related Side Effects and Adverse Reactions; Mild Cognitive Impairment; Breast Cancer
Keywords: Chemo-brain; Drug-Related Side Effects and Adverse Reactions; Mild Cognitive Impairment; Breast cancer
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Cognitive Dysfunction; Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comprehensive acupuncture (CAI) (Active Comparator): Breast cancer patients receiving Cytoxan-containing chemotherapy regimens (Chemo) will receive Dense cranial electroacupuncture stimulation (DCEAS) and Body acupuncture (BA).
  Interventions: Procedure: Dense cranial electroacupuncture stimulation; Procedure: Body acupuncture; Drug: Cytoxan-containing chemotherapy regimens
- Least acupuncture stimulation (LAS) (Sham Comparator): Breast cancer patients receiving Cytoxan-containing chemotherapy regimens (Chemo) will receive Least acupuncture stimulation (LAS)
  Interventions: Procedure: Least acupuncture stimulation; Drug: Cytoxan-containing chemotherapy regimens

INTERVENTIONS:
Procedure: Dense cranial electroacupuncture stimulation — DCEAS is a is a novel stimulation mode in which electrical stimulation is delivered on acupoints located on the forehead.
  Six pairs of acupoints are used: Baihui (GV20) and Yintang (EX-HN3), left Sishencong (EX-HN1) and Toulinqi (GB15), right Sishencong (EX-HN1) and Toulinqi (GB15), bilateral Shuaigu (GB8), bilateral Taiyang (EX-HN5), and bilateral Touwei (ST8).
  Disposable acupuncture needles (Hwato®, 0.30 mm in diameter and 25-40 mm in length) are inserted at a depth of 10-30 mm perpendicularly or obliquely into acupoints. Manual manipulation is then conducted to evoke needling sensation, followed by electrical stimulation (ITO ES-160, continuous waves at 2 Hz).
  Other Names: DCEAS
  Arms: Comprehensive acupuncture (CAI)
Procedure: Body acupuncture — Following acupoints are used: Shui-Gou (GV26), Shen-Men (HT7). He-Gu (LI4), Wai-Guan (TE5), Zhong-Wan (CV12), Guan-Yuan (CV4), Zu-San-Li (ST36), Feng-Long (ST40) and San-Yin-Jiao (SP6).
  Disposable acupuncture needles (Hwato®, 0.30 mm in diameter and 25-40 mm in length) are inserted at a depth of 10-30 mm perpendicularly or obliquely into acupoints. Manual manipulation is then conducted to evoke needling sensation. No electrical stimulation is delivered.
  Other Names: BA
  Arms: Comprehensive acupuncture (CAI)
Procedure: Least acupuncture stimulation — The acupoints chosen are less related to the treated syndromes based on Traditional Chinese Medicine (TCM) theory; the number of acupoints used and the intensity of electrical stimulation are also lower than the comprehensive acupuncture regimen. The following 6 acupoints will be used in LAS control: bilateral Tong-Tian (GB17), bilateral Shou San-Li (LI10) and bilateral Fu-Yang (BL59). Electrical stimulation will be only performed on bilateral Tong-Tian (GB17) and the intensities are adjusted to a level at which patients just start feeling the stimulation.
  Other Names: LAS
  Arms: Least acupuncture stimulation (LAS)
Drug: Cytoxan-containing chemotherapy regimens — Each subject shall receive oral administration or venous injection or both with adjuvant or neoadujuvant chemotherapy regimens, as decided by clinical oncologist.
  In clinical practice, the most commonly used Cytoxan-containing regimens include but are not limit to:
  AC (x4) [Adriamycin + Cytoxan], TC (x4) [Taxotere + Cytoxan], AC-P (4+4) [Adriamycin + Cytoxan + Paclitaxel], TAC (x6) [Taxotere + Adriamycin + Cytoxan], or AC-PH (4+4) [Adriamycin + Cytoxan + Paclitaxel + Herceptin].
  Other Names: Chemo

SUMMARY:
Chemobrain is an expression used to describe a cluster of chemotherapy-induced cognitive impairment symptoms, including problems with visual and verbal memory, forgetfulness, difficulty in learning, attention, concentration and coordination of multitasking and organization. Over 75% cancer patients experienced acute cognitive symptoms during chemotherapy and 17%-34% of them have long-term post-treatment cognitive deficits which can persist up to 10 years. Breast cancer survivors even display as high as 50%-75% prevalence of post-treatment cognitive impairment. Chemobrain has become an apparent quality-of-life issue for cancer survivors and will be encountered more frequently with the rise of the number of cancer survivors. There are no effective interventions available for preventing and treating chemobrain.

Acupuncture is beneficial in reducing various side effects of anti-cancer treatment. It also shows the efficacy in improving mild cognitive impairment and other dementia disorders; facilitates the recovery of pathological microstructural changes of the brain. These results have led to the hypothesis that acupuncture is effective in preventing chemobrain and this preventive effect may be associated with the protection against cytokine production, epigenetic modification and microstructural changes of the brain.

To test this hypothesis, an assessor-blinded, randomised controlled trial will be conducted to determine if a combination of DCEAS and body acupuncture could reduce the incidence and symptoms of chemobrain in breast cancer patients under chemotherapy compared to least acupuncture stimulation (LAS) as controls.

A total of 168 breast cancer patients who are ready for chemotherapy will be randomly assigned to comprehensive acupuncture intervention (combined DCEAS and body acupuncture regimen + chemotherapy) (CAI) (n = 84) for 2 sessions per week for 8 weeks or least acupuncture stimulation (LAS) (minimal acupuncture + chemotherapy) (n = 84). All patients receive the standard chemotherapy of breast cancer. Treatment outcomes on cognitive performance, fatigue and the depression will be assessed.

DETAILED DESCRIPTION:
Although the development of various chemotherapeutic drugs has greatly improved clinical outcomes and survival rate of cancer patients, it also causes various adverse side effects. Chemotherapy-induced cognitive impairment, often referred to as chemobrain, has drawn increasing attention due to the rise in the number of cancer survivors over the past decade. Numerous studies have shown that chemotherapy can cause acute and long-term post-treatment cognitive impairment, including problems with visual and verbal memory, forgetfulness, difficulty in learning, attention, concentration and coordination of multitasking and organization. Over 75% cancer patients reported to experience acute cognitive symptoms during chemotherapy and 17%-34% of them have long-term post-treatment cognitive deficits which can persist up to 10 years. Breast cancer survivors may display higher prevalence of post-treatment cognitive impairment. The severity of reported chemobrain symptoms is variable, from subtle to more severe. Chemobrain has become an apparent quality-of-life issue for survivors and will be encountered more frequency in the future. However, there are no effective interventions available to prevent and treat chemobrain, although some pharmacological, antioxidant and various cognitive approaches have been tested.

It is believed that chemobrain is a consequence of brain neuronal injury induced by systemically administered chemotherapeutic agents via direct and indirect mechanisms, resulting in the suppression of neuronal cell proliferation, epigenetic modification and microstructural changes of the brain. These pathological circumstances are largely developed from alternations in cytokine milieu. While physical and psychological stressors that cancer patients experienced after diagnosis, chemotherapy and long-term follow-up have been shown to increase circulating cytokine levels and increased cytokine levels are associated with cognitive decline in cancer patients, the administration of chemotherapy also results in cytokine production at peripheral and central levels as the medications induce tumor cell death and collateral tissue injury. Patients undergoing chemotherapy have been found to display significant increases in multiple cytokines.

A large body of evidence well confirms that acupuncture is effective in reducing anti-cancer treatment-caused side effects, including pain, nausea, hot flashes, fatigue, xerostomia, anxiety, depression and sleep disturbance. Numerous studies further have shown the effectiveness of acupuncture therapy in improving cognitive function of patients with mild cognitive impairment (MCI) and various dementia. The reduced severity of cognitive symptoms is associated with neuroimaging improvement in brain regions associated with learning and memory process. Acupuncture also ameliorates cognitive impairment in various animal models. Studies have further revealed that the cognition-improving effects of acupuncture are associated with the inhibition of cytokine-mediated neuronal cell apoptosis, inflammatory reaction and oxidative cellular injury and the effects in reducing cognitive symptoms are related to the protection of neuronal cells, improvement of electrophysiological activities of the hippocampus and brain cell proliferation. Moreover, acupuncture also displays a significant effect in facilitating the recovery of the brain at microstructural histopathological level in patients with cerebral infarction and in rats with transient focal cerebral ischemia. The investigators therefore hypothesize that acupuncture may be also effective in preventing and reducing chemotherapy caused cognitive impairment.

Recently, the investigators have developed a novel acupuncture stimulation called dense cranial electroacupuncture stimulation (DCEAS) on the basis of neuroanatomical rationale. In this mode, electrical stimulation is delivered on dense acupoints located on the forehead innervated by the trigeminal nerve. The trigeminal sensory pathway has much intimate fiber connections with brain regions associated with sensory, locomotor, visceral function, sleep, emotion, learning and memory. Therefore, DCEAS can effectively modulate brain functions. Over the past 5 years, the investigators have completed several clinical studies and demonstrated the benefits of DCEAS in the treatment of major depression, insomnia, OCD, postpartum depression and post-stroke depression. In the proposed study, a combination of DCEAS and body acupuncture will be employed to prevent and treat chemobrain in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese females aged 18 to 65 years;
2. have a diagnosis of stage I-IIIa breast cancer; and
3. are ready for orally administered or vein injection or both with Cytoxan-containing regimens as adjuvant chemotherapy before or after surgical treatment or in combination with other pharmacotherapy.

Exclusion Criteria:

1. had chemotherapy in the last 2 years;
2. have cardiac pacemakers, epilepsy or other unstable medical conditions;
3. had investigational drug treatment within the past 6 months;
4. alcoholism or drug abuse within the past 1 year; or
5. have severe needle phobia.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Changes in cognitive function (objective measurement) | Baseline, 2 week, 4 week, 6 week, 8 week
  The Montreal Cognitive Assessment (MoCA) of corresponding dialects will be used as an objective measurement for subjects' cognitive function. Assessments will be conducted at baseline and every 2 weeks thereafter.
Changes in cognitive function (subjective measurement) | Baseline, 2 week, 4 week, 6 week, 8 week
  The Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) of corresponding dialects will be used as a subjective measurement for subjects' cognitive function. Assessments will be conducted at baseline and every 2 weeks thereafter.

SECONDARY OUTCOMES:
Changes in quality of Life - composite measure | Baseline, 4 week, 8 week
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (QLQ-C30+BR23) and Functional Assessment of Cancer Therapy-Breast (FACT-B) of corresponding dialects will be used for assessment on quality of life. Both of them will be used as the former focuses on physical function, while the latter emphasizes on emotional well-being. Assessments will be conducted at baseline and every 4 weeks thereafter.
Changes in illness related fatigue measured by FACIT-Fatigue | Baseline, 4 week, 8 week
  As fatigue is a common co-morbidity observed in patients receiving chemotherapy, it will be measured using the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) of corresponding dialects. Assessments will be conducted at baseline and every 4 weeks thereafter.
Changes in chemo adverse effects - composite measure | Baseline, 4 week, 8 week
  Adverse side effects will be assessed using Functional Assessment of Cancer Therapy questionnaires (FACT-Taxane, FACT-BRM) of corresponding dialects. Assessments will be conducted at baseline and every 4 weeks thereafter.
Changes in subject perception of chemotherapy treatment measured by FACIT-TS-G | Baseline, 4 week, 8 week
  To determine whether acupuncture can reduce the adverse effects of chemo-therapy treatment and therefore increase subject acceptance, subject treatment satisfaction will be assessed using Functional Assessment of Chronic Illness Therapy questionnaire (FACIT-TS-G). Assessments will be conducted at baseline and every 4 weeks thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang-Jin ZHANG, MMed, PhD, Principal Investigator — School of Chinese Medicine, The University of Hong Kong
Locations (6):
- China (2):
  - Department of Chinese Medicine, The University of Hong Kong - Shenzhen Hospital, Shenzhen, Guangdong
  - Department of Clinical Oncology, The University of Hong Kong - Shenzhen Hospital, Shenzhen, Guangdong
- Hong Kong (4):
  - The Nethersole School of Nursing, The Chinese University of Hong Kong, Shatin, N.T.
  - Department of Clinical Oncology, Queen Mary Hospital, Hong Kong
  - Department of Surgery, Queen Mary Hospital, Hong Kong
  - Department of Surgery, Tung Wah Hospital, Sai Ying Pun

REFERENCES:
- [Background] Nelson CJ, Nandy N, Roth AJ. Chemotherapy and cognitive deficits: mechanisms, findings, and potential interventions. Palliat Support Care. 2007 Sep;5(3):273-80. doi: 10.1017/s1478951507000442. PMID 17969831
- [Background] Asher A. Cognitive dysfunction among cancer survivors. Am J Phys Med Rehabil. 2011 May;90(5 Suppl 1):S16-26. doi: 10.1097/PHM.0b013e31820be463. PMID 21765260
- [Background] Hede K. Chemobrain is real but may need new name. J Natl Cancer Inst. 2008 Feb 6;100(3):162-3, 169. doi: 10.1093/jnci/djn007. Epub 2008 Jan 29. No abstract available. PMID 18230787
- [Background] Matsuda T, Takayama T, Tashiro M, Nakamura Y, Ohashi Y, Shimozuma K. Mild cognitive impairment after adjuvant chemotherapy in breast cancer patients--evaluation of appropriate research design and methodology to measure symptoms. Breast Cancer. 2005;12(4):279-87. doi: 10.2325/jbcs.12.279. PMID 16286908
- [Background] Avisar A, River Y, Schiff E, Bar-Sela G, Steiner M, Ben-Arye E. Chemotherapy-related cognitive impairment: does integrating complementary medicine have something to add? Review of the literature. Breast Cancer Res Treat. 2012 Nov;136(1):1-7. doi: 10.1007/s10549-012-2211-5. Epub 2012 Aug 23. PMID 22915072
- [Background] Briones TL, Woods J. Chemotherapy-induced cognitive impairment is associated with decreases in cell proliferation and histone modifications. BMC Neurosci. 2011 Dec 9;12:124. doi: 10.1186/1471-2202-12-124. PMID 22152030
- [Background] Simo M, Rifa-Ros X, Rodriguez-Fornells A, Bruna J. Chemobrain: a systematic review of structural and functional neuroimaging studies. Neurosci Biobehav Rev. 2013 Sep;37(8):1311-21. doi: 10.1016/j.neubiorev.2013.04.015. Epub 2013 May 6. PMID 23660455
- [Background] Garcia MK, McQuade J, Haddad R, Patel S, Lee R, Yang P, Palmer JL, Cohen L. Systematic review of acupuncture in cancer care: a synthesis of the evidence. J Clin Oncol. 2013 Mar 1;31(7):952-60. doi: 10.1200/JCO.2012.43.5818. Epub 2013 Jan 22. PMID 23341529
- [Background] Chou P, Chu H, Lin JG. Effects of electroacupuncture treatment on impaired cognition and quality of life in Taiwanese stroke patients. J Altern Complement Med. 2009 Oct;15(10):1067-1073. PMID 20050300
- [Background] Guo Y, Shi X, Uchiyama H, Hasegawa A, Nakagawa Y, Tanaka M, Fukumoto I. A study on the rehabilitation of cognitive function and short-term memory in patients with Alzheimer's disease using transcutaneous electrical nerve stimulation. Front Med Biol Eng. 2002;11(4):237-47. doi: 10.1163/156855701321138905. PMID 12735425
- [Background] Yu J, Zhang X, Liu C, Meng Y, Han J. Effect of acupuncture treatment on vascular dementia. Neurol Res. 2006 Jan;28(1):97-103. doi: 10.1179/016164106X91951. PMID 16464371
- [Background] Zhao L, Zhang H, Zheng Z, Huang J. Electroacupuncture on the head points for improving gnosia in patients with vascular dementia. J Tradit Chin Med. 2009 Mar;29(1):29-34. doi: 10.1016/s0254-6272(09)60027-3. PMID 19514185
- [Background] Zhou Y, Jin J. Effect of acupuncture given at the HT 7, ST 36, ST 40 and KI 3 acupoints on various parts of the brains of Alzheimer' s disease patients. Acupunct Electrother Res. 2008;33(1-2):9-17. PMID 18672741
- [Background] Manni L, Aloe L, Fiore M. Changes in cognition induced by social isolation in the mouse are restored by electro-acupuncture. Physiol Behav. 2009 Dec 7;98(5):537-42. doi: 10.1016/j.physbeh.2009.08.011. Epub 2009 Sep 3. PMID 19733189
- [Background] Yu J, Liu C, Zhang X, Han J. Acupuncture improved cognitive impairment caused by multi-infarct dementia in rats. Physiol Behav. 2005 Nov 15;86(4):434-41. doi: 10.1016/j.physbeh.2005.07.015. Epub 2005 Sep 21. PMID 16181648
- [Background] Yu J, Yu T, Han J. Aging-related changes in the transcriptional profile of cerebrum in senescence-accelerated mouse (SAMP10) is remarkably retarded by acupuncture. Acupunct Electrother Res. 2005;30(1-2):27-42. doi: 10.3727/036012905815901370. PMID 16231630
- [Background] Cheng H, Yu J, Jiang Z, Zhang X, Liu C, Peng Y, Chen F, Qu Y, Jia Y, Tian Q, Xiao C, Chu Q, Nie K, Kan B, Hu X, Han J. Acupuncture improves cognitive deficits and regulates the brain cell proliferation of SAMP8 mice. Neurosci Lett. 2008 Feb 20;432(2):111-6. doi: 10.1016/j.neulet.2007.12.009. Epub 2007 Dec 15. PMID 18215464
- [Background] Shen Y, Li M, Wei R, Lou M. Effect of acupuncture therapy for postponing Wallerian degeneration of cerebral infarction as shown by diffusion tensor imaging. J Altern Complement Med. 2012 Dec;18(12):1154-60. doi: 10.1089/acm.2011.0493. Epub 2012 Sep 5. PMID 22950816
- [Background] Wu Z, Hu J, Du F, Zhou X, Xiang Q, Miao F. Long-term changes of diffusion tensor imaging and behavioural status after acupuncture treatment in rats with transient focal cerebral ischaemia. Acupunct Med. 2012 Dec;30(4):331-8. doi: 10.1136/acupmed-2012-010172. Epub 2012 Oct 16. PMID 23074236
- [Background] Zhang ZJ, Wang XM, McAlonan GM. Neural acupuncture unit: a new concept for interpreting effects and mechanisms of acupuncture. Evid Based Complement Alternat Med. 2012;2012:429412. doi: 10.1155/2012/429412. Epub 2012 Mar 8. PMID 22474503
- [Background] Zhang ZJ, Ng R, Man SC, Li TY, Wong W, Tan QR, Wong HK, Chung KF, Wong MT, Tsang WK, Yip KC, Ziea E, Wong VT. Dense cranial electroacupuncture stimulation for major depressive disorder--a single-blind, randomized, controlled study. PLoS One. 2012;7(1):e29651. doi: 10.1371/journal.pone.0029651. Epub 2012 Jan 6. PMID 22238631
- [Background] Zhang ZJ, Wang XY, Tan QR, Jin GX, Yao SM. Electroacupuncture for refractory obsessive-compulsive disorder: a pilot waitlist-controlled trial. J Nerv Ment Dis. 2009 Aug;197(8):619-22. doi: 10.1097/NMD.0b013e3181b05fd1. PMID 19684500
- [Background] Whitley E, Ball J. Statistics review 4: sample size calculations. Crit Care. 2002 Aug;6(4):335-41. doi: 10.1186/cc1521. Epub 2002 May 10. PMID 12225610
- [Background] Man SC, Hung BH, Ng RM, Yu XC, Cheung H, Fung MP, Li LS, Leung KP, Leung KP, Tsang KW, Ziea E, Wong VT, Zhang ZJ. A pilot controlled trial of a combination of dense cranial electroacupuncture stimulation and body acupuncture for post-stroke depression. BMC Complement Altern Med. 2014 Jul 19;14:255. doi: 10.1186/1472-6882-14-255. PMID 25038733
- [Background] Qu SS, Huang Y, Zhang ZJ, Chen JQ, Lin RY, Wang CQ, Li GL, Wong HK, Zhao CH, Pan JY, Guo SC, Zhang YC. A 6-week randomized controlled trial with 4-week follow-up of acupuncture combined with paroxetine in patients with major depressive disorder. J Psychiatr Res. 2013 Jun;47(6):726-32. doi: 10.1016/j.jpsychires.2013.02.004. Epub 2013 Mar 14. PMID 23498306
- [Background] Zhong LL, Tong Y, Tang GW, Zhang ZJ, Choi WK, Cheng KL, Sze SC, Wai K, Liu Q, Yu BX. A randomized, double-blind, controlled trial of a Chinese herbal formula (Er-Xian decoction) for menopausal symptoms in Hong Kong perimenopausal women. Menopause. 2013 Jul;20(7):767-76. doi: 10.1097/GME.0b013e31827cd3dd. PMID 23793167
- [Background] Han JS. Acupuncture: neuropeptide release produced by electrical stimulation of different frequencies. Trends Neurosci. 2003 Jan;26(1):17-22. doi: 10.1016/s0166-2236(02)00006-1. No abstract available. PMID 12495858
- [Background] Hammerschlag R. Methodological and ethical issues in clinical trials of acupuncture. J Altern Complement Med. 1998 Summer;4(2):159-71. doi: 10.1089/acm.1998.4.159. PMID 9628206
- [Background] Bergh J. Best use of adjuvant systemic therapies II, chemotherapy aspects: dose of chemotherapy-cytotoxicity, duration and responsiveness. Breast. 2003 Dec;12(6):529-37. doi: 10.1016/s0960-9776(03)00162-0. PMID 14659131
- [Background] Yeung PY, Wong LL, Chan CC, Leung JL, Yung CY. A validation study of the Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) in Chinese older adults in Hong Kong. Hong Kong Med J. 2014 Dec;20(6):504-10. doi: 10.12809/hkmj144219. Epub 2014 Aug 15. PMID 25125421
- [Background] Cheung YT, Lim SR, Shwe M, Tan YP, Chan A. Psychometric properties and measurement equivalence of the English and Chinese versions of the functional assessment of cancer therapy-cognitive in Asian patients with breast cancer. Value Health. 2013 Sep-Oct;16(6):1001-13. doi: 10.1016/j.jval.2013.06.017. PMID 24041350
- [Background] McLachlan SA, Devins GM, Goodwin PJ. Validation of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (QLQ-C30) as a measure of psychosocial function in breast cancer patients. Eur J Cancer. 1998 Mar;34(4):510-7. doi: 10.1016/s0959-8049(97)10076-4. PMID 9713301
- [Background] Schagen SB, Muller MJ, Boogerd W, Rosenbrand RM, van Rhijn D, Rodenhuis S, van Dam FS. Late effects of adjuvant chemotherapy on cognitive function: a follow-up study in breast cancer patients. Ann Oncol. 2002 Sep;13(9):1387-97. doi: 10.1093/annonc/mdf241. PMID 12196364
- [Background] Chie WC, Chang KJ, Huang CS, Kuo WH. Quality of life of breast cancer patients in Taiwan: validation of the Taiwan Chinese version of the EORTC QLQ-C30 and EORTC QLQ-BR23. Psychooncology. 2003 Oct-Nov;12(7):729-35. doi: 10.1002/pon.727. PMID 14502597
- [Background] Ng R, Lee CF, Wong NS, Luo N, Yap YS, Lo SK, Chia WK, Yee A, Krishna L, Goh C, Cheung YB. Measurement properties of the English and Chinese versions of the Functional Assessment of Cancer Therapy-Breast (FACT-B) in Asian breast cancer patients. Breast Cancer Res Treat. 2012 Jan;131(2):619-25. doi: 10.1007/s10549-011-1764-z. Epub 2011 Sep 16. PMID 21922244
- [Background] Nguyen J, Popovic M, Chow E, Cella D, Beaumont JL, Chu D, DiGiovanni J, Lam H, Pulenzas N, Bottomley A. EORTC QLQ-BR23 and FACT-B for the assessment of quality of life in patients with breast cancer: a literature review. J Comp Eff Res. 2015 Mar;4(2):157-66. doi: 10.2217/cer.14.76. PMID 25825844
- [Background] Wang SY, Zang XY, Liu JD, Gao M, Cheng M, Zhao Y. Psychometric properties of the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) in Chinese patients receiving maintenance dialysis. J Pain Symptom Manage. 2015 Jan;49(1):135-43. doi: 10.1016/j.jpainsymman.2014.04.011. Epub 2014 May 28. PMID 24878068
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Webster K, Cella D, Yost K. The Functional Assessment of Chronic Illness Therapy (FACIT) Measurement System: properties, applications, and interpretation. Health Qual Life Outcomes. 2003 Dec 16;1:79. doi: 10.1186/1477-7525-1-79. PMID 14678568
- [Derived] Zhang ZJ, Man SC, Yam LL, Yiu CY, Leung RC, Qin ZS, Chan KS, Lee VHF, Kwong A, Yeung WF, So WKW, Ho LM, Dong YY. Electroacupuncture trigeminal nerve stimulation plus body acupuncture for chemotherapy-induced cognitive impairment in breast cancer patients: An assessor-participant blinded, randomized controlled trial. Brain Behav Immun. 2020 Aug;88:88-96. doi: 10.1016/j.bbi.2020.04.035. Epub 2020 Apr 16. PMID 32305573